CLINICAL TRIAL: NCT06255886
Title: Treatment of Gastroesophageal Reflux Disease in Infants- a Randomized Controlled Trial
Brief Title: Treatment of Gastroesophageal Reflux Disease in Infants
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OUH-HCA006
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Gastroesophageal Reflux; Infant, Newborn, Diseases
Keywords: Reflux; Infants; GERD; GER; GORD; GOR; Cow milk protein; Bovine milk protein; CMP; Proton pump inhibitor; PPI; Omeprazole
MeSH Terms: conditions — Gastroesophageal Reflux; Infant, Newborn, Diseases | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is partially blinded. There is blinding in relation to the placebo arm and the proton pump inhibitor arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proton pump inhibitor (Active Comparator): Omeprazole 1 mg/ kg and continuing nutrition containing cow's milk protein
  Interventions: Drug: Protein pump inhibitor.
- Mother or infant diet (Active Comparator): Mother on cow milk-protein-free diet if breastfeeding and infant on a hypoallergenic formula if bottle-fed.
  Interventions: Behavioral: Mother or infant diet
- Placebo (Placebo Comparator): Placebo medicine (appearing substantially like Omeprazole) 1mg/kg and continuing nutrition containing cow's milk protein
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Protein pump inhibitor. — 1 mg/kg /day
  Other Names: Omeprazole
  Arms: Proton pump inhibitor
Behavioral: Mother or infant diet — Mother on cow milk protein diet or infant on hypoallergenic formula in case of bottle fed
  Other Names: Cow milk protein free diet
  Arms: Mother or infant diet
Drug: Placebo — Placebo medicine (appearing substantially like Omeprazole) 1mg/ ml, and continuing nutrition containing cows' milk protein
  Arms: Placebo

SUMMARY:
Gastroesophageal reflux disease in infants is not fully understood. Infants are prescribed medical treatments that may not be effective or that contribute to adverse side effects and lead to concerns and expenses for the parents and healthcare system. Current guidelines recommend cow-milk-protein free diet as a first-line treatment, but these recommendations are based on weak evidence. This study investigate the efficacy of a cow-milk-protein free diet compared to treatment with a proton pump inhibitor (omeprazole)

DETAILED DESCRIPTION:
An increasing number of infants less than one year of age have been referred to the pediatric departments with gastroesophageal reflux in the past decade. Gastroesophageal reflux is a common condition in infants defined as the passage of gastric contents into the esophagus with regurgitation or vomiting. Around 50% of infants younger than four months regurgitate or vomit regularly. In most cases, it is a harmless, self-limiting condition; in 90% of cases, the symptoms diminish before 12 months. However, if reflux leads to troublesome symptoms or complications, it is defined as gastroesophageal reflux disease. Troublesome symptoms may include failure to thrive, back arching, food refusal, regurgitation, and irritability. The prevalence of gastroesophageal reflux disease varies between studies. Infants can be treated medically, and proton pump Inhibitors have been recommended as the first choice. However, within the last few years, there has been concern among pediatricians that too many infants are unnecessarily treated with this medication. There are only a few randomized studies on proton pump inhibitor treatment in children under one year, and most studies do not show a significant effect on symptoms. Side effects of treatment with proton pump inhibitors include symptoms related to the gastrointestinal tract or airways, increased susceptibility to infections, and increased risk of developing allergy later in life. Within the past years, there has been attention to the overlapping of symptoms between gastroesophageal reflux disease and allergy to cow milk protein. Cow-milk-protein allergy is the most common food allergy in early childhood, with an estimated prevalence of 2-3%, and presents with various symptoms predominantly from the skin and gastrointestinal tract. Consequently, cow-milk-protein allergy can be challenging to differentiate from gastroesophageal reflux disease. Cow-milk-protein-allergy is an immune reaction and can be either immunoglobulin E-mediated, presenting with immediate reaction including anaphylaxis, or non-immunoglobulin E-mediated, presenting with delayed symptoms. In addition, it is possible that cow's milk can aggravate gastroesophageal reflux disease with a non-immunologic mechanism. As there is no biomarker to differentiate non-immunoglobulin E-mediated cow-milk allergy from gastroesophageal reflux disease, the diagnosis of non-immunoglobulin E-mediated cow-milk allergy can only be verified by an oral food challenge test preceded by a cow-milk-protein-elimination period. Therefore, in the updated international guidelines, all children with gastroesophageal reflux disease should start with a 2-4-week cow-milk-protein-elimination diet before a proton pump inhibitor is prescribed. However, evidence is scarce on the effect of a cow-milk-protein-free diet in infants diagnosed with gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with gastroesophageal reflux disease (GERD)
* Age < 1 year at the time of referral
* Age >1 month at start of treatment
* At least 3 reflux episodes/daily in average
* At least one of following troublesome symptoms are present: Crying of unknown reason, discomfort/irritability, problems gaining weight/ weightloss, rejects the breast or bottle, apnea, back-arching.

Exclusion Criteria:

* Children with diagnosed or suspected syndrome /genetic disorder
* Congenital malformations (minor deformities are excepted)
* Abdominal surgery
* Metabolic disease
* Treatment with proton pump inhibitor within the last week
* Allergy for proton pump inhibitors
* Allergy for cow milk protein
* Infants on Cow's milk free diet

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in reflux episodes in the fourth week of active treatment, compared to placebo | Baseline and daily in 4 weeks.
  Parent-reported reduction in the weekly number of reflux-episodes in the fourth week of active treatment with either PPI or diet, compared to placebo. The outcome is registered daily in an App.

SECONDARY OUTCOMES:
Change from baseline in reflux episodes in the fourth week in the PPI group, compared to the diet group. | Baseline and 4 weeks
  Reduction in the number of regurgitation episodes (compared to the run-in period) in the PPI group compared to the diet group
Change from baseline in weight | Baseline and 4 weeks
  A nurse or physician will perform the measurement on a weight in the clinic/hospital. Measurement unit: gram.
Change from baseline in the number of reflux episodes with visible blood | 1,2,3,4 weeks
  Parent reported weekly number of reflux episodes with visible blood. Registered in MyCap App.
Change from baseline in the number of episodes with discomfort | 1,2,3,4 weeks
  Parent reported weekly episodes with discomfort 5 minutes after feeding. Registered in MyCap App
Change from baseline in the numbers of episodes with crying | 1,2,3,4 weeks
  Parent reported weekly numbers of episodes with crying 5 minutes after feeding. Registered in MyCap App
Change from baseline in the number of episodes of refusing breast/ bottle | 1,2,3,4 weeks
  Parent reported weekly numbers of episodes of refusing breast/bottle. Registered in MyCap App
Change from baseline in the number of episodes with short breathing pauses | 1,2,3,4 weeks
  Parent-reported weekly numbers of episodes with short breathing pauses. Registered in MyCap App
Change from baseline in the number of episodes with paleness/blue color in face or lips | 1,2,3,4 weeks
  Parent reported weekly numbers of episodes with paleness/blue color in face. Registered in MyCap App
Change from baseline in the number of episodes with troublesome breathing/cough | 1,2,3,4 weeks
  Parent reported weekly numbers of episodes with troublesome breathing/cough. Registered in MyCap App
Immunoglobulin E level | 4 weeks after treatment is started
  Blood positive/negative for specific immunoglobulin E for cows milk protein. Values above 0,35 kU/l are considered positive for cows' milk allergy.

OTHER OUTCOMES:
Adverse events to trial medicine in the proton pump inhibitor group and the placebo group | 1,2,3,4 weeks
  Any parent-reported adverse events to the trial medicine (both Omeprazole and placebo) are registered weekly.
  There are several well-known side effects; 1-10 % experience symptoms from the gastrointestinal tract (i.e., stomach pain, nausea, and constipation), skin, airways, and increased susceptibility to infections.
Cows milk allergy? | 4 weeks
  After 4 weeks´ of cows milk protein-free diet, an oral provocation test with cow's milk is conducted on all infants in the diet group, who experienced effect of the diet. The test will be carried out in the hospital. During the test, the infants are given increasing doses of fresh cow's milk every 30 minutes until they reach a maximum of 200 ml.
  A nurse records any symptoms experienced during the first few hours of the test, and the parents are required to monitor and report any symptoms at home. Additionally, the parents inform the physician of any late symptoms via phone call 48 hours after the test.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Zachariassen, Professor, Study Director — H.C Andersen Childrens Hospital, Odense University Hospital and Syddansk University (SDU)
Locations (3):
- Denmark (3):
  - Paediatric Department, Hospital of Southern Jutland, Aabenraa, Region Syddanmark
  - Børnelægecentret v/Kasper Dalby, Odense, Region Syddanmark
  - H.C Andersen Childrens' Hospital, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No
Raw data can not be shared, but the study protocol and the Statistical Analysis plan will be shared.

REFERENCES:
- [Derived] Barkholt NK, Dalby K, Mogensen CB, Zachariassen G, Gradman J. Infant Reflux Trial: study protocol for a multicentre randomized controlled trial on the treatment of gastroesophageal reflux disease in infants. Trials. 2026 Jan 29. doi: 10.1186/s13063-026-09477-x. Online ahead of print. PMID 41612404